CLINICAL TRIAL: NCT02962609
Title: Comparing the Effect of Feeding Preterm Infants in Two Different Positions on Some Physiological Characteristics: A Randomized-Controlled Trial
Brief Title: Effect of Feeding Positions of Preterm Infants on Some Physiological Characteristics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, DUYGU GOZEN, Associate Professor of Nursing Faculty, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 48252- BAP IU
Record Dates: First submitted 2016-11-01; First posted 2016-11-11 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-09

CONDITIONS: Feeding Behavior
Keywords: Feeding; preterm infant; physiological characteristics; position; ESL; ESU
MeSH Terms: conditions — Feeding Behavior; Premature Birth

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Semielevated Side-Lying Position-ESL (Experimental): Preterm infants feed in the ESL position. In the ESL position, infant's head and trunk were elevated to an angle of 45-60° with the help of a pillow prepared by the researcher from the beds that were previously used in the unit and infants were held in side-lying position as in the breast-feeding position where their right ear faced the ceiling and the other ear faced the arms of the researcher. Their knees and hip were leaned against the researcher's arms and both the head and the neck were held at the same level by the researcher, whereas the chin was held in the flexion posture mildly facing the floor.
  Interventions: Other: Semielevated Side-lying Position-ESL
- Semielevated Supine Position-ESU (Experimental): Before feeding: In the ESU position, the head and the trunk of the infant were elevated to an angle of 45-60° with the help of the same pillow that was prepared by the researcher from the beds previously used in the unit and was used in the experimental group and the infant was laid in supine position in the arms of the researcher. Their head and neck were held at the same level by the researcher, whereas the chin was held in the flexion posture mildly facing the floor.
  Interventions: Other: Semielevated Supine Position

INTERVENTIONS:
Other: Semielevated Side-lying Position-ESL — The infants in the experimental group (n = 38) were held in the ESL position. In this position, their head and trunk were elevated to an angle of 45-60◦ with the help of a pillow prepared by the researcher from the beds that were previously used in the unit and infantswere held in the side-lying position as in the breast-feeding position where their right ear faced the ceiling and the other ear faced the arms of the researcher. Their knees and hip were leaned against the researcher's arms and their head and neck were held at the same level by the researcher; whereas, their chin was held in the flexion posture mildly facing the floor. The researcher supported their head, neck, and shoulder with her left hand and controlled the bottlewith her right hand.
  Arms: Semielevated Side-Lying Position-ESL
Other: Semielevated Supine Position — The ESU position was applied to the infants in the control group (n=42). In this position, their head and trunk were elevated to an angle of 45-60◦ with the help of the same pillow that was prepared by the researcher from the beds previously used in the unit and was used in the experimental group and they was laid in the supine position in the arms of the researcher. Their head and neck were held at the same level by the researcher, whereas their chin was held in the flexion posture mildly facing the floor. The researcher supported their head, neck, and shoulder with her left hand and controlled the bottlewith her right hand.
  Arms: Semielevated Supine Position-ESU

SUMMARY:
The purpose of this study is to determine the effect of Semielevated Side-Lying (ESL) and Semielevated Supine Position (ESU) positions used in bottle-feeding of very preterm infants upon their physiological characteristics and feeding performances.

DETAILED DESCRIPTION:
Semielevated supine position (ESU) is a position frequently used in neonatal intensive care units. In this position, infant is laid and fed on its back and the head is elevated to an angle of 45-60° in order to reduce the respiratory load of lungs. The ESL position, head of the infant is elevated to an angle of 45-60° and the infant is fed in the side-lying position. Since this position mimics the breast-feeding position, very preterm infants are supported to utilize the advantages of breast-feeding. A randomization was provided in the sample group consisting of totally 80 infants and while 38 infants were included in the ESL (experimental) group, 42 infants were included in the ESU (control) group.In the power analysis repeated at the end of the study, the power of the study was determined as 87% at a reliability of 95%.

ELIGIBILITY:
Inclusion Criteria:

* To be born between 26-31+6 gestational weeks according to mother's last menstruation date,
* To be between 32-39+6 postmenstrual weeks during the study,
* Have a body weight above 1500 g,
* Have a full enteral feeding,
* To be in a transition from orogastric catheter feeding to oral feeding for less than 24 hours,
* Have an oral feeding in this process for at least once,
* Tolerate at least 80% of amount of food given lastly during oral feeding,
* Voluntarily signing of the written informed consent form by parents

Exclusion Criteria:

* Infants suffering from craniofacial abnormalities like cleft palate,
* cleft lip and facial muscle paralysis; gastrointestinal, neurological and genetic disorders (necrotising enterocolitis, intracranial haemorrhage, periventricular leukomalacia, hydrocephalia, down syndrome, omphalocele, gastroschisis, short bowel syndrome etc.)
* moderate and severe bronchopulmonary dysplasia (BPD) (Jobe & Bancalari, 2001)
* patent ductus arteriosus requiring surgical therapy were excluded from the study

Ages: 32 Weeks to 38 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burcu AYKANAT GİRGİN, Principal Investigator — Istanbul University Florence Nightingale Faculty of Nursing

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Semielevated Side-Lying Position-ESL: Feeding Position. In the ESL position, infant's head and trunk were elevated to an angle of 45-60° with the help of a pillow prepared by the researcher from the beds that were previously used in the unit and infants were held in side-lying position as in the breast-feeding position where their right ear faced the ceiling and the other ear faced the arms of the researcher. Their knees and hip were leaned against the researcher's arms and both the head and the neck were held at the same level by the researcher, whereas the chin was held in the flexion posture mildly facing the floor.
  Feeding Position: Semielevated side-lying position (ESL): Experimental Group Semielevated supine position (ESU): Control Group
- Semielevated Supine Position-ESU: Feeding Position. In the ESU position, the head and the trunk of the infant were elevated to an angle of 45-60° with the help of the same pillow that was prepared by the researcher from the beds previously used in the unit and was used in the experimental group and the infant was laid in supine position in the arms of the researcher. Their head and neck were held at the same level by the researcher, whereas the chin was held in the flexion posture mildly facing the floor.
  Feeding Position: Semielevated side-lying position (ESL): Experimental Group Semielevated supine position (ESU): Control Group
Period: Overall Study
Arm/Group | Semielevated Side-Lying Position-ESL | Semielevated Supine Position-ESU
Started | 38 | 42
Completed | 38 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Semielevated Side-Lying Position-ESL | Semielevated Supine Position-ESU | Total
Number analyzed (Participants) | 38 | 42 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 38 | 42 | 80
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: postmenstural age (weeks)] | 34 (1) | 34 (1) | 34 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 19 | 20 | 39
Region of Enrollment [Number; unit: participants]
  Turkey | 38 | 42 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Oxygen Saturation
Description: Oxygen saturation were measured by using a pulse oximeter 2 min before the feeding, during the feeding and for 30 min after the feeding.
Time Frame: During feeding (maximum 30 min)
Measure: Mean (Standard Deviation); unit: SpO2%
Arm/Group | Semielevated Side-Lying Position-ESL | Semielevated Supine Position-ESU
Number analyzed (Participants) | 38 | 42
SpO2%
  2 min Before the feeding | 98.08 (1.6) | 98.09 (1.7)
  During feeding | 96.7 (2.5) | 93.4 (5.6)
  30 min after the feeding | 97.9 (1.7) | 96.7 (2.8)

2. Secondary Outcome: Heart Rate/Minute During Feeding
Description: Heart rate were measured by using a pulse oximeter 2 min before the feeding, during the feeding and for 30 min after the feeding. Feeding duration, feeding efficiency, and percentage of food intake were evaluated via a video during the feeding and recorded after the feeding.
Time Frame: During feeding (maximum 30 min)
Measure: Mean (Standard Deviation); unit: Beats per min
Arm/Group | Semielevated Side-Lying Position-ESL | Semielevated Supine Position-ESU
Number analyzed (Participants) | 38 | 42
Beats per min
  2 min Before the feeding | 151.1 (14.7) | 150.3 (18.6)
  During feeding | 155.8 (11.1) | 164.3 (6.0)
  30 min after the feeding | 150.5 (10.7) | 155.1 (13.6)

3. Other Pre Specified Outcome: Feeding Performances
Description: Feeding duration (minute)
Time Frame: during feeding (maximum 30 min)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Semielevated Side-Lying Position-ESL | Semielevated Supine Position-ESU
Number analyzed (Participants) | 38 | 42
minutes | 13 (5) | 15 (6)

ADVERSE EVENTS:
Time Frame: 30 minutes after feeding
Description: During the feeding, the infants in both groups were followed up in terms of their physiological-behavioral stress and fatigue symptoms in accordance with the cue-based feeding approach and the feeding was interrupted for a short time in case of these symptoms. The feeding was continued in case of the cues showing that they were ready to be fed again as well as physiological stability.
Arm/Group | Semielevated Side-Lying Position-ESL | Semielevated Supine Position-ESU
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/42
Other Adverse Events (participants affected / at risk) | 0/38 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
When the research is published, it has to describe that "this research is funded by Istanbul University Scientific Research Project"